CLINICAL TRIAL: NCT00952744
Title: Copeptin Helps in the Early Detection Of Patients With Acute Myocardial
Brief Title: Investigation of the Biomarker Copeptin in Patients With Acute Myocardial Infarction
Acronym: CHOPIN
Status: Completed | Type: Observational
Sponsor: Brahms AG (Industry)
Responsible Party: Sponsor
Other Study IDs: CHOPIN
Record Dates: First submitted 2009-07-20; First posted 2009-08-06 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Acute Coronary Syndromes
Keywords: acute myocardial infarction; ST-segment elevation myocardial infarction; STEMI; non-ST-segment elevation myocardial infarction; NSTEMI; unstable angina; unstable angina pectoris; UA; UAP
MeSH Terms: conditions — Acute Coronary Syndrome; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction; Angina, Unstable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples
Oversight: Data Monitoring Committee: No

SUMMARY:
While troponin is not detectable until several hours after an Acute Myocardial Infarction (AMI), copeptin is expected to be elevated very early after an AMI. A combination of both markers for the diagnosis of AMI early after the event is therefore expected to be advantageous.

DETAILED DESCRIPTION:
In patients with symptoms suggestive of acute coronary syndrome (ACS) such as chest pain or pressure, shortness of breath, diaphoresis, and nausea, detection of a rise and/or fall of troponin with at least one value above the 99th percentile of the upper reference limit is essential to the diagnosis of acute myocardial infarction (AMI). However, current troponin testing has limitations, including antibody specificity, assay imprecision, lack of standardization and a relatively late increase in the circulating troponin level after the onset of ischemia. Studies have shown a low diagnostic sensitivity of troponins when measured early (<6 hours) after symptom onset. Although there are some more sensitive troponin assays with a coefficient of variation (CV)10% at the 99th percentile of a normal reference population, most troponin assays have an imprecision CV of around 20% at the 99th percentile of the reference population. The early insensitivity of troponin results in an unmet need in the clinical evaluation of patients presenting with suspected ACS and AMI.

Copeptin may improve early AMI diagnostic sensitivity because of a number of unique characteristics.

* Copeptin levels are elevated at presentation in patients with AMI compared to patients with other presentations.
* Copeptin levels are elevated in patients with AMI even when troponin levels were not elevated at the time of initial presentation.
* Thus, a combination of troponin and copeptin levels at presentation may result in a more accurate diagnosis of acute AMI than troponin alone.
* Copeptin levels drop 1 day after an AMI.

ELIGIBILITY:
Inclusion Criteria:

* The subject must be 18 years of age or older.
* The subject must present to the Emergency Department with symptoms consistent with acute coronary syndromes (e.g., chest discomfort/pain, squeezing/fullness in the chest, pain radiating to left or both arms, jaw pain, pain in the back/neck/stomach, shortness of breath, cold sweat, nausea/vomiting, lightheadedness).
* The subject must present to the Emergency Department within 6 hours of the onset of the most recent symptoms that prompted the subject to seek medical attention in the Emergency Department.
* The patient agrees to abide by all aspects of the protocol, including all telephone follow-up.

Exclusion Criteria:

* The patient is unable to provide consent or understand the consent form.
* The ACS symptoms are clearly not the result of ACS (i.e., penetrating wounds, crush injury, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the ED with symptoms consistent with acute coronary syndromes.
Sampling Method: Probability Sample
Enrollment: 2071 (Actual)
Dates: Start 2009-08; Primary Completion 2010-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Copeptin improves early diagnostic performance for AMI when used in combination with troponin for the initial blood draw in patients presenting to the emergency department with symptoms consistent with acute coronary syndromes. | at initial presentation, at 2 hours, at 6 hours

SECONDARY OUTCOMES:
Copeptin improves AMI diag and is prog for outcome. Risk MACE > for 4th qrt. of MR-proADM than 1st. Copeptin adds to phys. assessment for AMI diag. Copeptin >18 pmol/l distinguishes between AMI and UA or other. Copeptin < 18 pmol/l excludes NSTEMI. | within 180 days after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Alan S Maisel, MD, Principal Investigator — Veteran's Affairs Medical Center San Diego, University of California San Diego; W Frank Peacock, MD, Study Chair — The Cleveland Clinic; Christian Mueller, MD, Study Chair — University Hospital, Basel, Switzerland
Locations (11):
- United States (11):
  - Stanford University Hospital, Palo Alto, California
  - University of California, San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Kansas University Medical Center, Kansas City, Kansas
  - University of Maryland, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - The Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Virginia Commonwealth University, Richmond, Virginia

REFERENCES:
- [Derived] Shah KS, Marston NA, Mueller C, Neath SX, Christenson RH, McCord J, Nowak RM, Vilke GM, Daniels LB, Hollander JE, Apple FS, Cannon CM, Nagurney J, Schreiber D, deFilippi C, Hogan CJ, Diercks DB, Limkakeng A, Anand IS, Wu AH, Clopton P, Jaffe AS, Peacock WF, Maisel AS. Midregional proadrenomedullin predicts mortality and major adverse cardiac events in patients presenting with chest pain: results from the CHOPIN trial. Acad Emerg Med. 2015 May;22(5):554-63. doi: 10.1111/acem.12649. Epub 2015 Apr 23. PMID 25908114
- [Derived] Maisel A, Mueller C, Neath SX, Christenson RH, Morgenthaler NG, McCord J, Nowak RM, Vilke G, Daniels LB, Hollander JE, Apple FS, Cannon C, Nagurney JT, Schreiber D, deFilippi C, Hogan C, Diercks DB, Stein JC, Headden G, Limkakeng AT Jr, Anand I, Wu AHB, Papassotiriou J, Hartmann O, Ebmeyer S, Clopton P, Jaffe AS, Peacock WF. Copeptin helps in the early detection of patients with acute myocardial infarction: primary results of the CHOPIN trial (Copeptin Helps in the early detection Of Patients with acute myocardial INfarction). J Am Coll Cardiol. 2013 Jul 9;62(2):150-160. doi: 10.1016/j.jacc.2013.04.011. Epub 2013 Apr 30. PMID 23643595